CLINICAL TRIAL: NCT03158311
Title: A Multicenter, Partially-Blinded, Randomized, 24-Week, Parallel-Group, Non-Inferiority, Open-Label Active Controlled Study to Compare the Efficacy and Safety of QVM149 With a Free Triple Combination of Salmeterol/Fluticasone + Tiotropium in Patients With Uncontrolled Asthma
Brief Title: Study to Compare QVM149 and Free Triple Combination of Salmeterol/Fluticasone + Tiotropium
Acronym: ARGON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CQVM149B2306; 2017-000136-34 (EudraCT Number)
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Results first posted 2020-10-14 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Asthma
Keywords: QVM149; Asthma; Moderate Asthma; Severe Asthma; ICS/LABA/LAMA; ICS/LABA; LAMA; Adult
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; Fluticasone; Tiotropium Bromide

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: The free triple combination of salmeterol/fluticasone + tiotropium was open label, for which investigators and patients had full knowledge that the patient had been assigned free triple combination comparator treatment. Within the two QVM149 treatment arms patients, investigator staff, and persons performing the assessments, remained blind to the identity of the actual QVM149 treatment dose but had full knowledge that the patient had been assigned QVM149 as study treatment. The data analysts and sponsor team were blinded to Case Report Forms that reveal the treatment arm. Randomization data and treatment codes were kept strictly confidential until the time of unblinding, and was not accessible by anyone else involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- QVM149 150/50/80 μg (Experimental): QVM149 150/50/80 μg o.d. delivered via Concept1
  Interventions: Drug: QVM149
- QVM149 150/50/160 μg (Experimental): QVM149 150/50/160 μg o.d. delivered via Concept1
  Interventions: Drug: QVM149
- Salmeterol/fluticasone 50/500 μg plus tiotropium 5 μg (Active Comparator): Salmeterol/fluticasone 50/500 μg b.i.d. delivered via Accuhaler® plus tiotropium 5 μg o.d. delivered via Respimat®
  Interventions: Drug: Salmeterol/fluticasone plus tiotropium

INTERVENTIONS:
Drug: QVM149 — Indacaterol acetate / glycopyrronium bromide / mometasone furoate
  Arms: QVM149 150/50/160 μg; QVM149 150/50/80 μg
Drug: Salmeterol/fluticasone plus tiotropium — Free triple arm of salmeterol / fluticasone plus tiotropium
  Arms: Salmeterol/fluticasone 50/500 μg plus tiotropium 5 μg

SUMMARY:
The purpose of this trial was to demonstrate that the efficacy of two treatment arms of the fixed-dose combination product QVM149 was non-inferior to the efficacy of the free combination arm of salmeterol/ fluticasone+ tiotropium in uncontrolled moderate to severe asthmatic patients.

The planned duration of treatment in this study was 24 weeks, followed up by a 7-day follow-up period.

DETAILED DESCRIPTION:
This study used a randomized, partially-blinded, 24-week, parallel-group, non-inferiority, open-label active controlled design. The study was partially open-label. Investigators and patients had knowledge of treatment allocation between QVM149 and/or comparator, however the QVM149 strength allocation was masked. The global sponsor team responsible for data review and analysis was blinded to all treatment allocations The study consisted of a screening period of up to 1-week, run-in period of 2-weeks, randomized treatment period of 24-weeks, and a follow-up period of 1-week.

At the screening visit, informed consent was obtained, and current and prohibited medications were reviewed. Rescue medication was provided to all patients who met the eligibility criteria and was to be used on an "as needed" basis throughout the study.

At the run-in visit, inclusion and exclusion criteria were reviewed and the patients were supplied with open-label long acting β2-adrenergic agonist/inhaled corticosteroids (LABA/ICS) salmeterol/fluticasone 50/250 μg b.i.d or 50/500 μg b.i.d to match their ICS background medication dose to be stopped at randomization visit.

All patients who met the eligibility criteria were randomized to 1 of 3 treatment arms with a randomization ratio of 1:1:1. The patients were stratified at randomization according to the ICS dose component of background ICS/LABA (medium or high dose) and region.

Treatment period visits were scheduled every 8 weeks. The study used two doses of QVM149 (high dose [150/50/160 μg] and a medium dose [150/50/80 μg] o.d. delivered via Concept1 inhaler) and a comparator treatment (salmeterol/fluticasone 50/500 μg b.i.d. delivered via Accuhaler® plus tiotropium 5 μg o.d delivered via Respimat®).

All randomized patients were contacted (by telephone) 7 days following the last dose of study medication or last visit, whichever was later, for Safety Follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of asthma for a period of at least 6 months prior to Visit 1 with current asthma severity ≥ step 4 (GINA 2017).
* Patients who had used ICS/LABA combinations for asthma for at least 3 months and at stable medium or high dose of ICS/LABA for at least 1 month prior to Visit 1.
* Patients were required to be symptomatic at screening despite treatment with medium or high stable doses of ICS/LABA as defined by ACQ-7 score ≥ 1.5 at visits 101 and 201 (randomization visit).
* Patients with history of at least one severe asthma exacerbation which required medical care from a physician, emergency room visit (or local equivalent structure) or hospitalization in the 12 months prior to Visit 1 and required systemic corticosteroid treatment for at least 3 days including physician guided self-management treatment with oral corticosteroids as part of written asthma action plan.
* Pre-bronchodilator FEV1 of < 85 % of the predicted normal value for the patient after withholding bronchodilators prior to spirometry at both Visit 101 and Visit 201.
* Patients who demonstrated an increase in FEV1 of ≥ 12% and 200 ml.

Exclusion Criteria:

* Patients who had a smoking history of greater than 20 pack years.
* Patients diagnosed with Chronic Obstructive Pulmonary Disease (COPD).
* Patients who had an asthma attack/exacerbation requiring systemic steroids or hospitalization or emergency room visit within 6 weeks of Visit 1 (Screening).
* Patients treated with a LAMA for asthma within 3 months prior to Visit 1.
* Patients who had a respiratory tract infection or clinical significant asthma worsening as defined by Investigator within 4 weeks prior to Visit 1 or between Visit 1 and Visit 201.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1426 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (121):
- Argentina (19):
  - Novartis Investigative Site, Berazategui, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Florida, Buenos Aires
  - Novartis Investigative Site, Lanús, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Nueve de Julio, Buenos Aires
  - Novartis Investigative Site, Ranelagh, Partido de Berazate, Buenos Aires
  - Novartis Investigative Site, Concepción del Uruguay, Entre Ríos Province
  - Novartis Investigative Site, Santa Rosa, La Pampa Province
  - Novartis Investigative Site, Buenos Aires, Nueve De Julio
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Bahía Blanca
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Salta
  - Novartis Investigative Site, Santa Fe
- Chile (2):
  - Novartis Investigative Site, Curicó, Maule Region
  - Novartis Investigative Site, Santiago, Santiago Metropolitan
- Colombia (2):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Bogotá
- Czechia (5):
  - Novartis Investigative Site, Ostrava Poruba, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Teplice, CZE
  - Novartis Investigative Site, Lovosice
  - Novartis Investigative Site, Miroslav
- Germany (24):
  - Novartis Investigative Site, Peine, Lower Saxony
  - Novartis Investigative Site, Geesthacht, Schleswig-Holstein
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Böhlen
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Einbeck
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Fürstenwalde
  - Novartis Investigative Site, Gelsenkirchen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Ludwigsburg
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Menden
  - Novartis Investigative Site, Mittweida
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Schleswig
  - Novartis Investigative Site, Witten
- Greece (3):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
- Hungary (8):
  - Novartis Investigative Site, Püspökladány, HUN
  - Novartis Investigative Site, Balassagyarmat
  - Novartis Investigative Site, Gödöllő
  - Novartis Investigative Site, Komló
  - Novartis Investigative Site, Sellye
  - Novartis Investigative Site, Siófok
  - Novartis Investigative Site, Szarvas
  - Novartis Investigative Site, Szeged
- India (9):
  - Novartis Investigative Site, Vijayawada, Andhra Pradesh
  - Novartis Investigative Site, Kozhikode, Kerala
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Mohali, Punjab
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Kolkata, West Bengal
- Israel (3):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
- Mexico (2):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
- Peru (4):
  - Novartis Investigative Site, San Martín de Porres, Lima region
  - Novartis Investigative Site, Santiago de Surco, Lima region
  - Novartis Investigative Site, Cusco
  - Novartis Investigative Site, Lima
- Poland (2):
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Poznan
- Russia (9):
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Ulyanovsk
  - Novartis Investigative Site, Yekaterinburg
- Serbia (4):
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Kamenitz
  - Novartis Investigative Site, Kragujevac
  - Novartis Investigative Site, Niš
- Slovakia (6):
  - Novartis Investigative Site, Bojnice, Slovak Republic
  - Novartis Investigative Site, Humenné, Slovak Republic
  - Novartis Investigative Site, Liptovský Hrádok, Slovak Republic
  - Novartis Investigative Site, Liptovský Mikuláš
  - Novartis Investigative Site, Topoľčany
  - Novartis Investigative Site, Žilina
- South Africa (5):
  - Novartis Investigative Site, Berea, Durban
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Chatsworth
  - Novartis Investigative Site, Kempton Park
  - Novartis Investigative Site, Pretoria
- Spain (5):
  - Novartis Investigative Site, Esparraguera, Barcelona
  - Novartis Investigative Site, Hostalets de Balenya, Catalonia
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, Benalmádena, Malaga
  - Novartis Investigative Site, Alzira, Valencia
- Taiwan (3):
  - Novartis Investigative Site, Kaoshiung, Taiwan
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Yenisehir/Izmir
- Vietnam (3):
  - Novartis Investigative Site, Ho Chi Minh City, VNM
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 166 investigative sites in 20 countries from 05 Feb 2018 to 19 Jul 2019.
Pre-assignment Details: A total of 1917 participants were screened. A 2 week run-in phase preceded the randomized treatment phase of the study. 1821 participants entered the run-in phase. Those participants who met the inclusion criteria entered the randomized treatment phase. Participants were randomized with a randomization ratio of 1:1:1 to three treatment arms.
Period: Overall Study
Arm/Group | QVM149 150/50/80 μg | QVM149 150/50/160 μg | Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg
Started (All participants who were assigned a randomization number) | 474 | 476 | 476
Full Analysis Set (FAS) (All the participants in the randomization set who received at least one dose of the study medication) | 474 | 476 | 475
Safety Set (SAF) (All the participants who received at least one dose of the study medication) | 474 | 476 | 475
Completed | 452 | 460 | 448
Not Completed | 22 | 16 | 28
Not completed — Subject/Guardian Decision | 10 | 6 | 11
Not completed — Adverse Event | 5 | 3 | 3
Not completed — Techinical Problems | 3 | 1 | 5
Not completed — Physician Decision | 2 | 3 | 7
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Sponsor decision | 1 | 0 | 0
Not completed — Pregnancy | 0 | 2 | 0
Not completed — Randomized in error | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QVM149 150/50/80 μg | QVM149 150/50/160 μg | Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg | Total
Number analyzed (Participants) | 474 | 476 | 476 | 1426
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.9 (13.58) | 52.7 (13.34) | 53.1 (13.08) | 52.5 (13.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 306 | 289 | 307 | 902
  Male | 168 | 187 | 169 | 524
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 10 | 16
  Asian | 36 | 34 | 33 | 103
  Black or African American | 6 | 5 | 3 | 14
  White | 401 | 392 | 391 | 1184
  Other | 26 | 44 | 39 | 109

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (AQLQ) Total Score
Description: The AQLQ is a 32-item asthma specific questionnaire designed to measure functional impairments that are most important to patients with asthma, with a recall time of two weeks and each question to be answered on a 7-point scale, where 1=totally limited/problems all the time and 7= not at all limited/no problems. It consists of 4 domains: symptoms, activity limitation, emotional funtion, and emotional stimuli. The overall score is calculated as the mean of 32 items. Higher AQLQ scores indicate better health-related quality of life.
Time Frame: Baseline and Week 24
Population: Analysis population included FAS with evaluable AQLQ data at both timepoints. No imputation was used for missing questions or missing total AQLQ score for this analysis. The analysis was performed on observed data only.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVM149 150/50/80 μg | QVM149 150/50/160 μg | Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg
Number analyzed (Participants) | 436 | 453 | 435
Score on a scale | 0.715 (0.070) | 0.827 (0.069) | 0.753 (0.069)
Statistical Analysis 1: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Test type: Non-Inferiority — Non-inferiority margin: 0.25 points; p < 0.001, Mixed Model for Repeated Measures (MMRM) — P-Value is one-sided; Least Square mean (LS Mean) = -0.038, 97.5% CI 1-sided [lower limit -0.139], Standard Error of Mean 0.051
Statistical Analysis 2: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Test type: Non-Inferiority — Non-inferiority margin: 0.25 points; p < 0.001, MMRM — P-Value is one-sided; LS Mean = 0.073, 97.5% CI 1-sided [lower limit -0.027], Standard Error of Mean 0.051

2. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. Trough FEV1 is the mean of two FEV1 values measures taken 15 minutes (min) and 45 min prior to evening dose.
Time Frame: Baseline, Week 8, Week 16 and Week 24
Population: Analysis population included FAS with FEV1 data at the respective visit. Number analyzed signified number of participants who were evaluable for this outcome measure at specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: Litre (L)
Arm/Group | QVM149 150/50/80 μg | QVM149 150/50/160 μg | Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg
Number analyzed (Participants) | 420 | 438 | 425
Litre (L)
  Week 8: number analyzed (Participants) | 382 | 395 | 371
  Week 8 | 0.246 (0.020) | 0.309 (0.020) | 0.243 (0.020)
  Week 16: number analyzed (Participants) | 357 | 389 | 371
  Week 16 | 0.251 (0.020) | 0.319 (0.020) | 0.253 (0.020)
  Week 24: number analyzed (Participants) | 367 | 385 | 372
  Week 24 | 0.248 (0.021) | 0.334 (0.021) | 0.238 (0.021)
Statistical Analysis 1: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 8; Test type: Superiority; p = 0.892, MMRM — P-value is two-sided; LS Mean = 0.003, 95% CI 2-sided [-0.046 to 0.052], Standard Error of Mean 0.025
Statistical Analysis 2: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 8; Test type: Superiority; p = 0.007, MMRM — P-value is two-sided; LS Mean = 0.067, 95% CI 2-sided [0.018 to 0.115], Standard Error of Mean 0.025
Statistical Analysis 3: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 16; Test type: Superiority; p = 0.945, MMRM — P-value is two-sided; LS Mean = -0.002, 95% CI 2-sided [-0.050 to 0.047], Standard Error of Mean 0.025
Statistical Analysis 4: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 16; Test type: Superiority; p = 0.007, MMRM — P-value is two-sided; LS Mean = 0.066, 95% CI 2-sided [0.018 to 0.114], Standard Error of Mean 0.025
Statistical Analysis 5: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 24; Test type: Superiority; p = 0.713, MMRM — P-value is two-sided; LS Mean = 0.009, 95% CI 2-sided [-0.041 to 0.060], Standard Error of Mean 0.026
Statistical Analysis 6: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 24; Test type: Superiority; p < 0.001, MMRM — P-value is two-sided; LS Mean = 0.096, 95% CI 2-sided [0.046 to 0.146], Standard Error of Mean 0.026

3. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ-7) Total Score
Description: The ACQ-7 measured asthma symptom control and consists of 7 items: 5 on symptom assessment, 1 on rescue medication use and 1 on airway calibre (FEV1 % predicted). All seven items are scored on a 7-point Likert scale, with 0 indicating total control and 6 indicating poor control. The questions are equally weighted and the total score is the mean of the seven items. Higher score indicates worst symptoms. The first 6 questions of the ACQ-7 were completed by the participant while the last question was completed by the study investigator using data from the Master Scope spirometer. A negative change from baseline indicates improvement in lung function.
Time Frame: Baseline, Week 16 and Week 24
Population: Analysis population included FAS with ACQ-7 data at the respective visit. Number analyzed signified number of participants who were evaluable for this measure at specified timepoints. No imputation was used for missing questions or missing total ACQ-7 score for this analysis. The analysis was performed on observed data only
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVM149 150/50/80 μg | QVM149 150/50/160 μg | Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg
Number analyzed (Participants) | 447 | 454 | 447
Score on a scale
  Week 16: number analyzed (Participants) | 436 | 441 | 428
  Week 16 | -1.043 (0.045) | -1.098 (0.045) | -1.020 (0.045)
  Week 24: number analyzed (Participants) | 437 | 452 | 436
  Week 24 | -1.080 (0.046) | -1.172 (0.045) | -1.048 (0.046)
Statistical Analysis 1: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 16; Test type: Superiority; p = 0.308, MMRM — P-value is one-sided; LS Mean = -0.023, 95% CI 2-sided [-0.113 to 0.067], Standard Error of Mean 0.046
Statistical Analysis 2: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 16; Test type: Superiority; p = 0.044, MMRM — P-value is one-sided; LS Mean = -0.079, 95% CI 2-sided [-0.169 to 0.012], Standard Error of Mean 0.046
Statistical Analysis 3: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 24; Test type: Superiority; p = 0.245, MMRM — P-value is one sided; LS Mean = -0.032, 95% CI 2-sided [-0.125 to 0.060], Standard Error of Mean 0.047
Statistical Analysis 4: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 24; Test type: Superiority; p = 0.004, MMRM — P-value is one sided; LS Mean = -0.124, 95% CI 2-sided [-0.216 to -0.032], Standard Error of Mean 0.047

4. Secondary Outcome: Change From Baseline in AQLQ Total Score
Description: The AQLQ is a 32-item asthma specific questionnaire designed to measure functional impairments that are most important to patients with asthma, with a recall time of two weeks and each question to be answered on a 7-point scale, where 1=totally limited/problems all the time and 7= not at all limited/no problems. It consists of 4 domains: symptoms, activity limitation, emotional function and environmental stimuli. The overall score is calculated as the mean of 32 items. Higher AQLQ scores indicate better health-related quality of life.
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVM149 150/50/80 μg | QVM149 150/50/160 μg | Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg
Number analyzed (Participants) | 435 | 442 | 429
Score on a scale | 0.690 (0.069) | 0.755 (0.068) | 0.673 (0.069)
Statistical Analysis 1: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Test type: Superiority; p = 0.719, MMRM — P-value is two-sided; LS Mean = 0.018, 95% CI 2-sided [-0.079 to 0.115], Standard Error of Mean 0.049
Statistical Analysis 2: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Test type: Superiority; p = 0.097, MMRM — P-value is two-sided; LS Mean = 0.082, 95% CI 2-sided [-0.015 to 0.179], Standard Error of Mean 0.049

5. Secondary Outcome: Percentage of Patients Achieving the Minimally Clinically Important Difference (MCID) Decrease From Baseline ACQ-7 ≥ 0.5
Description: The ACQ-7 measured asthma symptom control and consists of 7 items: 5 on symptom assessment, 1 on rescue medication use and 1 on airway calibre (FEV1 % predicted). All seven items are scored on a 7-point Likert scale, with 0 indicating total control and 6 indicating poor control. The questions are equally weighted and the total score is the mean of the seven items. Higher score indicates worst symptoms. The first 6 questions of the ACQ-7 were completed by the participant while the last question was completed by the study investigator using data from the Master Scope spirometer. A negative change from baseline indicates improvement in lung function. Decrease of ACQ-7 score of at least 0.5 from baseline was considered clinically meaningful.
Time Frame: Baseline and Week 24
Population: Analysis population included FAS with evaluable ACQ-7 data at both timepoints. Missing data imputation was used to perform this analysis. Subjects with missing values were imputed as non-responders (a non-responder was defined as <0.5 decrease in ACQ-7 score at week 24)
Measure: Count of Participants; unit: Participants
Arm/Group | QVM149 150/50/80 μg | QVM149 150/50/160 μg | Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg
Number analyzed (Participants) | 447 | 454 | 447
Participants | 393 | 387 | 375
Statistical Analysis 1: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Test type: Superiority; p = 0.061, Regression, Logistic — P-value is one sided; Logistic Regression Model via Generalized estimating equations (GEE); Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.94 to 1.61]
Statistical Analysis 2: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Test type: Superiority; p = 0.227, Regression, Logistic — P-value is one-sided; Logistic Regression Model via GEE; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.85 to 1.46]

6. Secondary Outcome: Percentage of Patients Achieving the Minimally Clinically Important Difference (MCID) Change From Baseline AQLQ ≥ 0.5
Description: The AQLQ is a 32-item asthma specific questionnaire designed to measure functional impairments that are most important to patients with asthma, with a recall time of two weeks and each question to be answered on a 7-point scale, where 1=totally limited/problems all the time and 7= not at all limited/no problems. It consists of 4 domains: symptoms, activity limitation, emotional function and environmental stimuli. The overall score is calculated as the mean of 32 items. Higher AQLQ scores indicate better health-related quality of life. An improvement of 0.5 points in AQLQ score is considered to be the minimally clinically important difference in asthma.
Time Frame: Baseline and Week 24
Population: Analysis population included FAS with evaluable AQLQ data at both timepoints. Missing data imputation was used to perform this analysis. Subjects with missing values were imputed as non-responders (a non-responder was defined as <0.5 increase in AQLQ score at week 24)
Measure: Count of Participants; unit: Participants
Arm/Group | QVM149 150/50/80 μg | QVM149 150/50/160 μg | Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg
Number analyzed (Participants) | 444 | 454 | 441
Participants | 318 | 333 | 299
Statistical Analysis 1: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Test type: Superiority; p = 0.108, Regression, Logistic — P-value is one sided; Logistic regression model via the GEE; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.91 to 1.49]
Statistical Analysis 2: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Test type: Superiority; p = 0.013, Regression, Logistic — P-Value is one sided; Logistic regression model via the GEE; Odds Ratio (OR) = 1.33, 95% CI 2-sided [1.03 to 1.70]

7. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: FVC is the total volume of air exhaled during a expiratory maneuvre. It was assessed by performing a spirometry assessment.
Time Frame: Baseline, Week 8, Week 16 and Week 24
Population: Analysis population included FAS with FVC data at the respective visit. Number analyzed signified number of participants who were evaluable for this measure at specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: Litre (L)
Arm/Group | QVM149 150/50/80 μg | QVM149 150/50/160 μg | Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg
Number analyzed (Participants) | 420 | 438 | 425
Litre (L)
  Week 8: number analyzed (Participants) | 382 | 395 | 371
  Week 8 | 0.216 (0.021) | 0.272 (0.021) | 0.219 (0.021)
  Week 16: number analyzed (Participants) | 357 | 389 | 371
  Week 16 | 0.221 (0.021) | 0.275 (0.021) | 0.217 (0.021)
  Week 24: number analyzed (Participants) | 367 | 385 | 372
  Week 24 | 0.214 (0.022) | 0.280 (0.022) | 0.186 (0.022)
Statistical Analysis 1: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 8; Test type: Superiority; p = 0.908, MMRM — P-Value is two-sided; LS Mean = -0.003, 95% CI 2-sided [-0.055 to 0.049], Standard Error of Mean 0.027
Statistical Analysis 2: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 8; Test type: Superiority; p = 0.046, MMRM — P-Value is two-sided; LS Mean = 0.053, 95% CI 2-sided [0.001 to 0.104], Standard Error of Mean 0.026
Statistical Analysis 3: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 16; Test type: Superiority; p = 0.870, MMRM — P-Value is two-sided; LS Mean = 0.004, 95% CI 2-sided [-0.047 to 0.056], Standard Error of Mean 0.026
Statistical Analysis 4: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 16; Test type: Superiority; p = 0.028, MMRM — P-Value is two-sided; LS Mean = 0.058, 95% CI 2-sided [0.006 to 0.109], Standard Error of Mean 0.026
Statistical Analysis 5: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 24; Test type: Superiority; p = 0.303, MMRM — P-Value is two-sided; LS Mean = 0.028, 95% CI 2-sided [-0.026 to 0.083], Standard Error of Mean 0.028
Statistical Analysis 6: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 24; Test type: Superiority; p < 0.001, MMRM — P-Value is two-sided; LS Mean = 0.095, 95% CI 2-sided [0.041 to 0.148], Standard Error of Mean 0.027

8. Secondary Outcome: Change From Baseline in Forced Expiratory Flow Between 25% and 75% of Forced Vital Capacity (FEF25-75)
Description: Forced expiratory flow during the mid (25 - 75%) portion of the FVC. It was assessed by performing spirometric assessment.
Time Frame: Baseline, Week 8, Week 16 and Week 24
Population: Analysis population included FAS with FEF25-75 data at the respective visit. Number analyzed signified number of participants who were evaluable for this measure at specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: Litres/second (L/s)
Arm/Group | QVM149 150/50/80 μg | QVM149 150/50/160 μg | Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg
Number analyzed (Participants) | 420 | 438 | 425
Litres/second (L/s)
  Week 8: number analyzed (Participants) | 382 | 395 | 371
  Week 8 | 0.290 (0.027) | 0.332 (0.027) | 0.270 (0.027)
  Week 16: number analyzed (Participants) | 357 | 389 | 371
  Week 16 | 0.291 (0.028) | 0.355 (0.027) | 0.297 (0.027)
  Week 24: number analyzed (Participants) | 367 | 385 | 372
  Week 24 | 0.290 (0.028) | 0.375 (0.028) | 0.286 (0.028)
Statistical Analysis 1: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 8; Test type: Superiority; p = 0.563, MMRM — P-value is two-sided; LS Mean = 0.020, 95% CI 2-sided [-0.048 to 0.087], Standard Error of Mean 0.034
Statistical Analysis 2: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 8; Test type: Superiority; p = 0.068, MMRM — P-Value is two-sided; LS Mean = 0.062, 95% CI 2-sided [-0.005 to 0.129], Standard Error of Mean 0.034
Statistical Analysis 3: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 16; Test type: Superiority; p = 0.844, MMRM — P-Value is two-sided; LS Mean = -0.007, 95% CI 2-sided [-0.076 to 0.062], Standard Error of Mean 0.035
Statistical Analysis 4: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 16; Test type: Superiority; p = 0.097, MMRM — P-Value is two-sided; LS Mean = 0.058, 95% CI 2-sided [-0.010 to 0.125], Standard Error of Mean 0.035
Statistical Analysis 5: Comparison: QVM149 150/50/80 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 24; Test type: Superiority; p = 0.927, MMRM — P-Value is two-sided; LS Mean = 0.003, 95% CI 2-sided [-0.067 to 0.074], Standard Error of Mean 0.036
Statistical Analysis 6: Comparison: QVM149 150/50/160 μg vs Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg; Week 24; Test type: Superiority; p = 0.013, MMRM — P-Value is two-sided; LS Mean = 0.089, 95% CI 2-sided [0.019 to 0.159], Standard Error of Mean 0.036

ADVERSE EVENTS:
Time Frame: Adverse events were collected starting on or after the time of first administration of study drug but not later than 7 days (30 days in case of a Serious Adverse Events) after the last administration, up to maximum duration of 203 days.
Description: Any sign or symptom that occurs during the study treatment but not later than 7 days (30 days in case of a Serious Adverse Events) after the last administration.
  Analysis performed on the safety set population. Safety Set consisted of all participants who received at least one dose of study medication during this study.
Groups:
- QVM149 150/50/80 μg: QVM149 150/50/80 µg o.d. delivered via Concept1
- QVM149 150/50/160 µg: QVM149 150/50/160 μg o.d. delivered via Concept1
Arm/Group | QVM149 150/50/80 μg | QVM149 150/50/160 µg | Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg
All-Cause Mortality (participants affected / at risk) | 0/474 | 0/476 | 1/475
Serious Adverse Events (participants affected / at risk) | 14/474 | 18/476 | 19/475
Other Adverse Events (participants affected / at risk) | 245/474 | 246/476 | 241/475
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVM149 150/50/80 μg (N=474) | QVM149 150/50/160 µg (N=476) | Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg (N=475)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Hyperpyrexia (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 5 | 0
Postoperative abscess (Infections and infestations) | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intentional product misuse (Injury, poisoning and procedural complications) | 0 | 0 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVM149 150/50/80 μg (N=474) | QVM149 150/50/160 µg (N=476) | Salmeterol/Fluticasone 50/500 μg Plus Tiotropium 5 μg (N=475)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 2 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0
Thyroid cyst (Endocrine disorders) | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 2
Eye disorder (Eye disorders) | 1 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0
Maculopathy (Eye disorders) | 0 | 0 | 1
Panophthalmitis (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 4
Dry mouth (Gastrointestinal disorders) | 3 | 1 | 5
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 4 | 4 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 2 | 0
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 7 | 3 | 4
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 1 | 1
Chills (General disorders) | 1 | 0 | 0
Discomfort (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Hyperpyrexia (General disorders) | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 0
Inflammation (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1
Pain (General disorders) | 0 | 1 | 0
Procedural failure (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 3 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 1
Atopy (Immune system disorders) | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 1
Perennial allergy (Immune system disorders) | 0 | 1 | 0
Abscess limb (Infections and infestations) | 2 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 2 | 3
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 21 | 22 | 19
Candida infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Chronic hepatitis C (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 2 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Ear infection fungal (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 2 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 5 | 3
Gingivitis (Infections and infestations) | 0 | 1 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 1 | 1
Infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 9 | 5 | 4
Laryngitis (Infections and infestations) | 3 | 3 | 2
Laryngitis viral (Infections and infestations) | 1 | 1 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 6 | 6 | 7
Nasopharyngitis (Infections and infestations) | 34 | 34 | 43
Oral candidiasis (Infections and infestations) | 1 | 2 | 4
Oral herpes (Infections and infestations) | 2 | 2 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 2 | 0 | 0
Perichondritis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 18 | 17 | 10
Pharyngitis bacterial (Infections and infestations) | 1 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 2
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 6 | 2 | 3
Respiratory tract infection viral (Infections and infestations) | 10 | 9 | 6
Rhinitis (Infections and infestations) | 7 | 5 | 4
Sinobronchitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 4 | 8 | 9
Skin infection (Infections and infestations) | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 3 | 3
Tonsillitis bacterial (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 1 | 1
Tracheitis (Infections and infestations) | 4 | 1 | 6
Tracheobronchitis (Infections and infestations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 13 | 10 | 9
Upper respiratory tract infection bacterial (Infections and infestations) | 5 | 9 | 9
Urinary tract infection (Infections and infestations) | 6 | 5 | 4
Viral infection (Infections and infestations) | 1 | 1 | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 1
Viral rhinitis (Infections and infestations) | 0 | 1 | 0
Viral tracheitis (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 8 | 11 | 10
Vulvovaginal candidiasis (Infections and infestations) | 1 | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Bronchial injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 4 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Exposure to allergen (Injury, poisoning and procedural complications) | 9 | 3 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 3 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 1
Breath sounds abnormal (Investigations) | 0 | 0 | 1
Crystal urine (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Haemoglobin increased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Liver function test increased (Investigations) | 1 | 0 | 0
Red blood cells urine (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Mineral metabolism disorder (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoporosis postmenopausal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 1
Convulsions local (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 10 | 15 | 9
Hemianopia (Nervous system disorders) | 0 | 0 | 1
Hypersomnia (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 4
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 0
Neuritis (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0
Phantom limb syndrome (Nervous system disorders) | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 2 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Tension headache (Nervous system disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 3 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 1
Pyelocaliectasis (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Breast disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 125 | 114 | 125
Catarrh (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Larynx irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 7 | 5 | 5
Malignant hypertension (Vascular disorders) | 1 | 0 | 0
Peripheral venous disease (Vascular disorders) | 1 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1
Varicophlebitis (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT03158311/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT03158311/SAP_001.pdf